CLINICAL TRIAL: NCT00877578
Title: Efficacy of a Special Oral Nutritional Supplement on Nutritional Status of Malnourished Elderly Patients
Acronym: Nutri-PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007/023/HP
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Malnutrition
Keywords: elderly patient; malnutrition; new nutritional support; micronutrients; elderly patient malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nutri-Energie ®, a cake of high caloric density and palatability, twice a day for 4 weeks, in addition to an enriched diet.
  Interventions: Dietary Supplement: Nutri-Energie ®, Aliscience society
- 2 (Active Comparator): Clinutren 1.5 ® standard isocaloric commercially available supplement, twice a day for 4 weeks, in addition to an enriched diet.
  Interventions: Dietary Supplement: Clinutren 1.5 ®, Nestlé Clinical Nutrition

INTERVENTIONS:
Dietary Supplement: Nutri-Energie ®, Aliscience society — Nutri-Energie ® is a new cake of high caloric density and palatability, enriched in different specific pharmaco nutrients.
  Arms: 1
Dietary Supplement: Clinutren 1.5 ®, Nestlé Clinical Nutrition — Clinutren 1.5 ®, isocaloric commercially available supplement, twice a day for 4 weeks, in addition to an enriched diet
  Arms: 2

SUMMARY:
The aim of this study is to evaluate in malnourished elderly patients the nutritional efficacy of a new nutritional supplement enriched in different specific pharmaco nutrients (leucine, micronutrients, omega-3) appearing in the form of a cake of high caloric density and palatability.

The primary endpoint is the outcome of fat-free mass measured by multiple frequence bio-impedance analysis.

DETAILED DESCRIPTION:
Ageing of the population and loss of autonomy expose to major consequences in terms of treatment charges and need for hospitalisation. Malnutrition has a key prognostic value, that worsen the prognosis of the primary disease; the length of hospital stay and the incidence of complications are related to nutritional status (Correia 2003, Pichard 2004, Schneider 2004). Several large scale studies at Rouen University Hospital, in 1998 and 2001, have revealed on more than 1000 patients (mid age 71 years) that malnutrition prevalence ranged of 35 to 38%, one third of which is severe (Jusserand 2000, Delaire 2002). Malnutrition increases the risk of complications (Naber 1997, Correia 2003), including muscle mass depletion, decrease of immune function and delayed wound healing. The main consequence of malnutrition is increased infectious morbidity and post operative mortality for the weakest patients. Increased length of hospital stay and rehabilitation duration also results in increased medicals and social burden, in particular in the elderly patients.

Recent studies have shown that usual hospital food intake was insufficient to cover patient's needs (Hébuterne 2001, Dupertuis 2003, Petit 2004) and that systematic nutritional screening was mandatory in hospitalised patients, using validated criteria and scales (e.g. NutriSteps®, MNA®).

The strategy for nutritional support includes as a first step enriched diets and the use of oral supplements, then enteral nutrition or even parenteral nutrition in the most severe cases (HAS guidelines 2007). The efficacy of oral supplementation has been proven (Stratton 2007). Yet, their composition still need to be optimised to better match specific nutritional needs and to ameliorate palatability and favour compliance.

The provision of specifics nutrients with anabolic, anti-oxidants or anti-inflammatory effects can optimise oral nutritional supplements, to achieve a true pharmaco-nutritional therapy. Accordingly, leucine enrichment has inhibitory effects on proteasome-mediated muscular proteolysis in aged rats (Combaret 2005). Trace elements deficiency (zinc, selenium, chromium, iron) is common in the elderly patients and increase the risk of infectious or wound complications (HAS 2007), and the level of trace elements provision in standard supplements may be insufficient to compensate this deficiency. Finally, omega-3 fatty acids enrichment enables to limit the inflammatory response and hypercatabolism (Delarue 2005).

The aim of this study is to evaluate in malnourished elderly patients the nutritional efficacy of a new nutritional supplement enriched in different specific pharmaco nutrients (leucine, micronutrients, omega-3) appearing in the form of a cake of high caloric density and palatability.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants
* Moderately malnourished defined by whether:

  18 < BMI < 21

  5 to 10% body weight loss in the last past 6 months.

Buzby index between 83.5 and 97.5 (calculated with weight loss and albumin)

* With or without any factors increasing malnutrition (insufficient caloric intakes, long term treatment)
* Justifying hospitalisation in rehabilitation unit

Exclusion Criteria:

* Age < 70 years old or > 90 years old
* Surgical affection involving a surgery in the next 10 days
* Contraindicated oral intakes due to digestive injury
* Total parenteral nutrition
* Ulcer or infection existing
* Malignant hemopathy
* Hepatic insufficiency (TP < 30%)
* Swallowing difficulties limiting solid oral intakes
* Kidney failure (renal dialysis)
* Expected survival > 3 months
* Impossibility to give an informed consent

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
outcome of fat-free mass measured by multiple frequence bio-impedance analysis | 28 days

SECONDARY OUTCOMES:
safety of oral supplementation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DECHELOTTE, PR, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Centre Hospitalier de Dieppe, Dieppe
  - UHRouen, Rouen